CLINICAL TRIAL: NCT05001035
Title: Effect of Different Biomimetic Materials on White Spot Lesions in Enamel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Eptesam Atef, Dental specialist at benha teaching hospital, Benha University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OP-P-018-001; OPDEN-107-1-G (Other: Faculty of dentistry Alazhar University girls branch)
Record Dates: First submitted 2021-07-28; First posted 2021-08-11 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: White Spot Lesion

STUDY DESIGN:
Intervention Model Description: Split mouth technique
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Zinc carbonated hydroxy apatite (Experimental): Toothpaste to be added on white spot lesions in dental enamel
  Interventions: Other: Time of assessment
- Bioactive glass (Experimental): Toothpaste to be added on white spot lesions in dental enamel
  Interventions: Other: Time of assessment
- Poly amido amine (Experimental): Resinous material to be painted on white spot lesions in dental enamel
  Interventions: Other: Time of assessment
- Control (No Intervention): No material to be added

INTERVENTIONS:
Other: Time of assessment — Immediate and after one month and after two months
  Arms: Bioactive glass; Poly amido amine; Zinc carbonated hydroxy apatite

SUMMARY:
This study will be conducted to evaluate: 1- The remineralizing effect of different biomimetic materials (Zinc carbonate hydroxyapatite nanoparticles, Poly-amido amine (PAMAM) and bioactive glass nanoparticles) on white spot lesions in enamel. 2- The clinical efficacy of these agents on disappearance of these white spots.

ELIGIBILITY:
Inclusion Criteria:

* Total of 21 patients enrolled in this study will be selected having at least 4 teeth (one on each quadrant) which will be extracted for orthodontic treatment.
* These patients will be selected according to age groups between 15-25 years old
* good oral hygiene
* free of destroying habits for dental tissues

Exclusion Criteria:

* Bruxism
* soft drinks consumption
* acid regurgitation, etc.).
* Selected teeth having any cracks, malformations, dysplasia or caries.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
change in remineralization from base line to time limit | Immediate and one month and two months
  Change in its density in digital xray
changes of appearance from base line photograph to time limit | Immediate and one month and two months
  White spots disappear on digital photography

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dental medicine for girls branch of Alazhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided